CLINICAL TRIAL: NCT06435975
Title: Pilot Study of Physical Activity Intervention to Manage Bowel Dysfunction in Rectal Cancer Survivors
Brief Title: Physical Activity in Rectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Erica Pettke, MD, MPH, FACS, Physician, Abramson Cancer Center at Penn Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 20221; 849585 (Other: Abramson Cancer Center of the University of Pennsylvania)
Record Dates: First submitted 2024-05-06; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Rectal Cancer; Rectosigmoid Cancer
Keywords: Rectal Cancer; Physical Activity; Bowel Dysfunction; Telehealth
MeSH Terms: conditions — Rectal Neoplasms; Motor Activity; Intestinal Diseases | interventions — Exercise; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Participants in this arm will be asked to complete a series of surveys, participate in telehealth-based interventions, and engage in moderate physical activity.
  Interventions: Other: Physical Activity; Other: Survey; Behavioral: Telehealth Lifestyle Coaching

INTERVENTIONS:
Other: Physical Activity — Participants will perform a baseline +4000 steps/day for the duration of the study. Aerobic exercise, similar to a brisk walk, will be recommended as the primary mode of exercise.
Other: Survey — Participants will complete a series of survey at multiple points throughout this study to assess quality of life issues. Questionnaires may be completed via paper forms with prepaid postage envelopes or using a REDCap online survey.
Behavioral: Telehealth Lifestyle Coaching — Participants will meet with a health coach, the Principal Investigator, to review baseline bowel habits and symptoms as well as discuss physical activity and potential strategies to achieve this goal, on a weekly basis for 12 weeks.

SUMMARY:
The goal of this clinical trial is to test a telehealth-based personalized physical activity intervention in adult patients diagnosed with Stage I-III rectal cancer. The main question it aims to answer are how to better understand the experiences of rectal cancer survivors who are coping with bowel dysfunction and how physical activity can improve their quality of life.

Participants will be asked to:

1. Complete surveys to assess bowel function and quality of life
2. Participate in 12 Telehealth Sessions (one session a week) to discuss and review bowel dysfunction
3. Perform daily physical activity

DETAILED DESCRIPTION:
The goal of this clinical trial is to administer and determine the feasibility of a personalized physical activity intervention for rectal cancer survivors. Structured physical activity interventions will be administered over a three-month period. An exit interview will be conducted at the completion of this time period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Stage I-III cancers of the rectum/rectosigmoid.
2. Age 18 or older
3. Three months to 5 years post-treatment completion
4. Have a rectal or anal anastomosis with a LARS score of 21-42
5. At least 10 participants must be racial/ethnic minority (Black/African American, Hispanic/Latino)
6. Ability to be physically active and cleared by MD
7. Patients must be able to read and understand English.
8. Participants must sign the informed consent form

The study is open to anyone regardless of gender or ethnicity. Efforts will be made to extend the accrual to a representative population, but in a trial which will accrue 20 subjects, a balance must be struck between subject safety considerations and limitations on the number of individuals exposed to potentially toxic or ineffective treatments on the one hand and the need to explore gender, racial, and ethnic aspects of clinical research on the other. If differences in outcome that correlate to gender, racial, or ethnic identity are noted, accrual may be expanded, or additional studies may be performed to investigate those differences more fully.

Exclusion Criteria:

1. Patients failing to meet all the above inclusion criteria will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of Physical Activity Intervention | From enrollment to the end of treatment at 12 weeks.
  Administer and determine the feasibility of a PA intervention. We will administer a telehealth physical activity intervention to 20 RC survivors (10 males and 10 females, at least 10 of which will be racial and/or ethnic minorities) over 12 weeks. Feasibility of the intervention will be measured by the percentage of participants who agree to participate of the total approached as well as completion of the intervention which will be defined as completion of ≥80% of the intervention (telehealth calls).

SECONDARY OUTCOMES:
Acceptability and Participant Satisfaction with Physical Activity Intervention | From enrollment to the end of treatment after 12 weeks.
  Using qualitative methods, evaluate the acceptability of and satisfaction with the intervention as reported by survivors. After completion of the intervention or decision to discontinue participation, we will administer a semi-structured exit interview to evaluate the acceptability of the intervention.
Evaluation using Memorial Sloan Kettering Cancer Center Bowel Function Instrument Scale to describe the change in total bowel symptom score in the pilot cohort from minimum score of 13 to maximum score of 65, where the higher score is the better outcome. | At 0 weeks, 3 weeks, and 6 months after completion of the initial intervention.
  Using the Memorial Sloan Kettering bowel function instrument administered pre-post PA intervention, describe the change in total bowel symptom score in the pilot cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Pettke, MD, MPH, FACS, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Hendren SK, O'Connor BI, Liu M, Asano T, Cohen Z, Swallow CJ, Macrae HM, Gryfe R, McLeod RS. Prevalence of male and female sexual dysfunction is high following surgery for rectal cancer. Ann Surg. 2005 Aug;242(2):212-23. doi: 10.1097/01.sla.0000171299.43954.ce. PMID 16041212
- [Background] Lange MM, van de Velde CJ. Urinary and sexual dysfunction after rectal cancer treatment. Nat Rev Urol. 2011 Jan;8(1):51-7. doi: 10.1038/nrurol.2010.206. Epub 2010 Dec 7. PMID 21135876
- [Background] Bruheim K, Guren MG, Skovlund E, Hjermstad MJ, Dahl O, Frykholm G, Carlsen E, Tveit KM. Late side effects and quality of life after radiotherapy for rectal cancer. Int J Radiat Oncol Biol Phys. 2010 Mar 15;76(4):1005-11. doi: 10.1016/j.ijrobp.2009.03.010. Epub 2009 Jun 18. PMID 19540058
- [Background] Hoerske C, Weber K, Goehl J, Hohenberger W, Merkel S. Long-term outcomes and quality of life after rectal carcinoma surgery. Br J Surg. 2010 Aug;97(8):1295-303. doi: 10.1002/bjs.7105. PMID 20602501
- [Background] Sun V, Grant M, Wendel CS, McMullen CK, Bulkley JE, Altschuler A, Ramirez M, Baldwin CM, Herrinton LJ, Hornbrook MC, Krouse RS. Dietary and Behavioral Adjustments to Manage Bowel Dysfunction After Surgery in Long-Term Colorectal Cancer Survivors. Ann Surg Oncol. 2015 Dec;22(13):4317-24. doi: 10.1245/s10434-015-4731-9. Epub 2015 Jul 10. PMID 26159443
- [Background] Krouse RS, Wendel CS, Garcia DO, Grant M, Temple LKF, Going SB, Hornbrook MC, Bulkley JE, McMullen CK, Herrinton LJ. Physical activity, bowel function, and quality of life among rectal cancer survivors. Qual Life Res. 2017 Nov;26(11):3131-3142. doi: 10.1007/s11136-017-1641-2. Epub 2017 Jul 4. PMID 28677077
- [Background] Fong DY, Ho JW, Hui BP, Lee AM, Macfarlane DJ, Leung SS, Cerin E, Chan WY, Leung IP, Lam SH, Taylor AJ, Cheng KK. Physical activity for cancer survivors: meta-analysis of randomised controlled trials. BMJ. 2012 Jan 30;344:e70. doi: 10.1136/bmj.e70. PMID 22294757
- [Background] Denlinger CS, Engstrom PF. Colorectal cancer survivorship: movement matters. Cancer Prev Res (Phila). 2011 Apr;4(4):502-11. doi: 10.1158/1940-6207.CAPR-11-0098. PMID 21464030
- [Background] Rock CL, Doyle C, Demark-Wahnefried W, Meyerhardt J, Courneya KS, Schwartz AL, Bandera EV, Hamilton KK, Grant B, McCullough M, Byers T, Gansler T. Nutrition and physical activity guidelines for cancer survivors. CA Cancer J Clin. 2012 Jul-Aug;62(4):243-74. doi: 10.3322/caac.21142. Epub 2012 Apr 26. PMID 22539238
- [Background] Grimmett C, Bridgewater J, Steptoe A, Wardle J. Lifestyle and quality of life in colorectal cancer survivors. Qual Life Res. 2011 Oct;20(8):1237-45. doi: 10.1007/s11136-011-9855-1. Epub 2011 Feb 1. PMID 21286822
- [Background] Brown JC, Schmitz KH. The prescription or proscription of exercise in colorectal cancer care. Med Sci Sports Exerc. 2014 Dec;46(12):2202-9. doi: 10.1249/MSS.0000000000000355. PMID 24781887
- [Background] Kushi LH, Doyle C, McCullough M, Rock CL, Demark-Wahnefried W, Bandera EV, Gapstur S, Patel AV, Andrews K, Gansler T; American Cancer Society 2010 Nutrition and Physical Activity Guidelines Advisory Committee. American Cancer Society Guidelines on nutrition and physical activity for cancer prevention: reducing the risk of cancer with healthy food choices and physical activity. CA Cancer J Clin. 2012 Jan-Feb;62(1):30-67. doi: 10.3322/caac.20140. PMID 22237782
- [Background] Ottenbacher A, Yu M, Moser RP, Phillips SM, Alfano C, Perna FM. Population Estimates of Meeting Strength Training and Aerobic Guidelines, by Gender and Cancer Survivorship Status: Findings From the Health Information National Trends Survey (HINTS). J Phys Act Health. 2015 May;12(5):675-9. doi: 10.1123/jpah.2014-0003. Epub 2014 May 15. PMID 24834485
- [Background] Bellizzi KM, Rowland JH, Jeffery DD, McNeel T. Health behaviors of cancer survivors: examining opportunities for cancer control intervention. J Clin Oncol. 2005 Dec 1;23(34):8884-93. doi: 10.1200/JCO.2005.02.2343. PMID 16314649
- [Background] Courneya KS, Katzmarzyk PT, Bacon E. Physical activity and obesity in Canadian cancer survivors: population-based estimates from the 2005 Canadian Community Health Survey. Cancer. 2008 Jun;112(11):2475-82. doi: 10.1002/cncr.23455. PMID 18428195
- [Background] Strid H, Simren M, Storsrud S, Stotzer PO, Sadik R. Effect of heavy exercise on gastrointestinal transit in endurance athletes. Scand J Gastroenterol. 2011 Jun;46(6):673-7. doi: 10.3109/00365521.2011.558110. Epub 2011 Mar 2. PMID 21366388
- [Background] Loprinzi PD, Lee H. Rationale for promoting physical activity among cancer survivors: literature review and epidemiologic examination. Oncol Nurs Forum. 2014 Mar 1;41(2):117-25. doi: 10.1188/14.ONF.117-125. PMID 24578072
- [Background] Schmitz KH, Holtzman J, Courneya KS, Masse LC, Duval S, Kane R. Controlled physical activity trials in cancer survivors: a systematic review and meta-analysis. Cancer Epidemiol Biomarkers Prev. 2005 Jul;14(7):1588-95. doi: 10.1158/1055-9965.EPI-04-0703. PMID 16030088
- [Background] Dainese R, Serra J, Azpiroz F, Malagelada JR. Effects of physical activity on intestinal gas transit and evacuation in healthy subjects. Am J Med. 2004 Apr 15;116(8):536-9. doi: 10.1016/j.amjmed.2003.12.018. PMID 15063815
- [Background] Hawkes AL, Chambers SK, Pakenham KI, Patrao TA, Baade PD, Lynch BM, Aitken JF, Meng X, Courneya KS. Effects of a telephone-delivered multiple health behavior change intervention (CanChange) on health and behavioral outcomes in survivors of colorectal cancer: a randomized controlled trial. J Clin Oncol. 2013 Jun 20;31(18):2313-21. doi: 10.1200/JCO.2012.45.5873. Epub 2013 May 20. PMID 23690410
- [Background] Hawkes AL, Pakenham KI, Courneya KS, Gollschewski S, Baade P, Gordon LG, Lynch BM, Aitken JF, Chambers SK. A randomised controlled trial of a tele-based lifestyle intervention for colorectal cancer survivors ('CanChange'): study protocol. BMC Cancer. 2009 Aug 18;9:286. doi: 10.1186/1471-2407-9-286. PMID 19689801
- [Background] Jonk Y, Lawson K, O'Connor H, Riise KS, Eisenberg D, Dowd B, Kreitzer MJ. How effective is health coaching in reducing health services expenditures? Med Care. 2015 Feb;53(2):133-40. doi: 10.1097/MLR.0000000000000287. PMID 25588134
- [Background] Goss F, Robertson R, DaSilva S, Suminski R, Kang J, Metz K. Ratings of perceived exertion and energy expenditure during light to moderate activity. Percept Mot Skills. 2003 Jun;96(3 Pt 1):739-47. doi: 10.2466/pms.2003.96.3.739. PMID 12831247
- [Background] Pearson ES. Goal setting as a health behavior change strategy in overweight and obese adults: a systematic literature review examining intervention components. Patient Educ Couns. 2012 Apr;87(1):32-42. doi: 10.1016/j.pec.2011.07.018. Epub 2011 Aug 17. PMID 21852063
- [Background] Demark-Wahnefried W, Rogers LQ, Alfano CM, Thomson CA, Courneya KS, Meyerhardt JA, Stout NL, Kvale E, Ganzer H, Ligibel JA. Practical clinical interventions for diet, physical activity, and weight control in cancer survivors. CA Cancer J Clin. 2015 May-Jun;65(3):167-89. doi: 10.3322/caac.21265. Epub 2015 Feb 13. PMID 25683894
- [Derived] Nehemiah A, Pettke EN, Appel S, Garcia DO, Bea JW, Thomson CA, Sun V, Krouse RS. Pilot Feasibility Study of Physical Activity to Manage Bowel Dysfunction in Survivors of Rectal Cancer. Dis Colon Rectum. 2025 Apr 1;68(4):483-490. doi: 10.1097/DCR.0000000000003583. Epub 2024 Dec 23. PMID 39714033
- See also: American Cancer Society. Cancer Facts & Figures 2020 — https://www.cancer.org/cancer/colon-rectal-cancer/about/key-statistics.html
- See also: 2018 Physical Activity Guidelines for Americans. US Department of Health and Human Services; 2008 — https://health.gov/sites/default/files/2019-09/Physical_Activity_Guidelines_2nd_edition.pdf